CLINICAL TRIAL: NCT05631834
Title: Bilateral Asymmetrical Erector Spinae Catheters Analgesia Versus Thoracic Epidural Catheter Analgesia in Minimally Invasive Oesophageal Cancer Surgery: a Randomized Controlled Trial
Brief Title: ESP Versus TEA for Oeasophagus Cancer Surgery
Acronym: ESPOK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vinmec Healthcare System (Other)
Responsible Party: Principal Investigator, Philippe Macaire, Director of anesthesia, Vinmec Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESP Oesophagus K
Record Dates: First submitted 2022-11-11; First posted 2022-11-30 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Peri Operative Analgesia

STUDY DESIGN:
Intervention Model Description: This is a single centered, open label, randomized controlled trial
Who Masked: Participant
Masking Description: This is a single centered, open label, randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Peri operative Thoracic epidural catheters analgesia (Active Comparator): Epidural catheter insertion will be performed at level T9 with catheter tip at level T7 After negative test dose with Lidocaine 2%, loading dose using Ropivacaine 0.5% (see table).
  Patient height (cm) Volume of LA (mL) 140-149 8 150-159 10 160-169 12 170-180 14 >180 16 Evaluation of sensory block should be at level T4 to T10 by cold test and pinprick. If extension needed, bolus of ropivacaine 0.5% 2 mL may be added.
  In post operative period▪ analgesia with intermitent automatic bolus UAB of ropivacaine 0.2% will be connected and started at 10 min after arrival in post operative care unit
  ▪ Pump preparation and settings: Patient 140 - 149 cm = 8 mL Patient 150 - 159 cm = 10 mL Patient 160 - 169 cm = 12 mL Patient 170 - 180 cm = 14 mL Patient >180 cm = 16 mL IAB every 4h reduced to 3h if needed Catheter will be removed 72h after end of surgery
  Interventions: Procedure: Thoracic epidurale
- Continuous Peri operative Bilateral erector spinae catheters analgesia (Experimental): The ESP will be performed Right side level The tip of the catheter should be on t T7.
  Left side level The tip of the catheter should be on T8.
  Induction with ropivacaine 0.5% with loading dose as follows:
  Patient height (cm) Volume of LA (mL) LEFT RIGHT 140-149 8 6 150-159 10 8 160-169 12 10 170-180 14 12 >180 16 14
  For post operative analgesia:
  * Pumps with intermittent automatic bolus (IAB) of ropivacaine 0.2% started at 10 min after arrival in PACU
  * Patient 140 - 149 cm = 6 mL / left side - 8 mL / right side
  * Patient 150 - 159 cm = 8 mL / left side - 10 mL / right side
  * Patient 160 - 169 cm = 10 mL / left side - 12 mL / right side
  * Patient 170 - 179 = 12 mL / left side - 14 mL / right side
  * Patient > 180 kg = 14 mL / side - 16 mL / right side The bolus on the second catheter will be delayed by 1 hour IAB every 6h Catheter will be removed 72h after end of surgery
  Interventions: Procedure: Erector spinae block

INTERVENTIONS:
Procedure: Thoracic epidurale — Epidurale Perioperative infusion of Ropivacaine
  Arms: Continuous Peri operative Thoracic epidural catheters analgesia
Procedure: Erector spinae block — erector spinae interfascia Perioperative infusion of Ropivacaine
  Arms: Continuous Peri operative Bilateral erector spinae catheters analgesia

SUMMARY:
For esophagectomy, peri-operative continuous thoracic epidural analgesia (TEA) is the standard of care for perioperative pain management. Although effective, TEA is associated with moderate to serious adverse events such as hypotension and neurologic complications. Peri-operative continuous Erector spinae analgesia (ESP) may be a safe alternative. The Investigators hypothesize that TEA and ESP are similar in efficacy for pain treatment in thoracolaparoscopic esophagectomy with less side effects.

Methods. This Randomized prospective randomized study will compare TEA (Which is a wellknown technique of regional anaesthesia with numerous publications) with ESP ( Which is a technique of regional anaesthesia described in 2016 and with already 1000 publication) in a consecutive series of 50 thoracolaparoscopic esophagectomies randomized in 2 groups study groups ESP and controled group TEA.

In this study,

* The TEA will consist of continuous epidural ropivacaine and sufen- tanil infusion with an induction dose for the surgery and a programmed intermittent bolus (PIB) started at the end of the surgery and ended 72h after the end of the surgery.
* The ESP; the Bilateral catheters will be inserted under ultrasound guidance after the anaesthesia induction with an induction dose and a PIB started at the end of the surgery and ended 72h after the end of the surgery.

The primary outcome will be the median highest recorded Visual Analogic Scale (VAS) during the 3 days after surgery.

The secondary outcomes will be vaso-pressor consumption, fluid administration, and length of hospital stay.

DETAILED DESCRIPTION:
For this single-center Prospective randomized controlled study, with the Approval of Ethical committee of VinMec Healthcare and after Patient's information waived the need for informed consent. The performance and reporting of this study will be in accordance with the Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) guidelines.

Investigators are hypothesizing that intra-operative and post operative Thoracic Epidural analgesia (TEA) or Erector Spinae Plane analgesia (ESP) are similary effective with regard to quality of analgesia in Thoraco Laparoscopic Akiyama oesophagectomy for cancer.

Patients, listed for this type of surgery,after information and signed consent will be randomized via a random number generator into one of two treatment groups by the person who obtained consent which is prescribed in the nurse preparation file".

• Group 1 = Control group will have peri-operative analgesia by standard Continuous TEA. The TEA performance and epidural insertion will be performed just before the anesthesia induction as per guidelines in regional anesthesia. the tip of the epidural cathter should be at the level of the thoracic vertebra (T) 7. Puncture point at level T9

Volume of ropivacaine 0.5% Patient height:

140 - 149 cm = 8 mL 150 - 159 cm = 10 mL 160 - 169 cm = 12 mL 170 - 180 cm = 14 mL >180 cm = 16 mL without exceeding 3 mg/kg

• Group 2 = Treatment group with have perioperative analgesia by continuous Bilateral ESP catheters. As it is interfascia block the guidelines of regional anesthesia allows to perform under general anesthesia (GA) The ESP performance will be just after inducation of GA on a stable patient. The ESP Performance performance will be under Ultrasound guidance. The tip of catheter will be on the left side at T6 and right side at T7.

Volume of ropivacaine 0.5% Patient height without exceeding 3 mg/kg 140 - 149 cm = 8 mL / left side - 6 mL / right side 150 - 159 cm = 10 mL / left side - 8 mL / right side 160 - 169 cm = 120 mL / left side - 10 mL / right side 170 - 179 cm= 14 mL / left side - 12 mL / right side > 180 cm = 16 mL / side - 14 mL / right side

After the surgery the patient will be extubated as soon as possible in the operating room and transferred to the intensive care unit for closed monitoring the post operative analgesia will Combined:

1. Paracetamol 15 mg/kg/dose every 8 h
2. Regional analgesia Ropivacaine 0,2% without exceeding 8mg/kg-24h. Group 1 TEA PIB every 4 hours 140 - 149 cm = 8 mL 150 - 159 cm = 10 mL 160 - 169 cm = 12 mL 170 - 180 cm = 14 mL >180 cm = 16 mL Group 2 ESP 140 - 149 cm = 8 mL / left side - 6 mL / right side 150 - 159 cm = 10 mL / left side - 8 mL / right side 160 - 169 cm = 120 mL / left side - 10 mL / right side 170 - 179 cm= 14 mL / left side - 12 mL / right side > 180 cm = 16 mL / side - 14 mL / right side
3. PCA morphine connected to the patient

   * Concentration Morphine : 50 mg/49 ml + Ketamine 50 mg
   * Loading dose: 1mg
   * PCA dose demand: 1 mL/dose
   * Lockout: 10 min
   * Continuous rate (basal): 0
   * Dose limit (hr): 6mg/hour Regional analgesia will be interrupted 72h after the induction of general anesthesia Analgesia will be

     * Paracetamol 500 mg x 3/day (Maximum 15mg/kg x 3 /day)
     * Arcoxia 60 mg BD
     * If pain = Ultracet maximum 3 per day

Control of plasmatic dosage ropivacaine 24h 48h 72h after induction ESP and 40 minutes after last PIB

Data collection will start just after induction of regional anaesthesia for both group up to 72h after the induction of the general anaesthesia

Statistical analysis The study is a non-inferiority trial. Two groups of patients scheduled for thoracoscopic oesophagectomy and receiving a TEA or ESP regional analgesia regimen were randomized and compared. As a non-inferiority trial, a per protocol analysis is mandatory. We consider that a patient non receiving a regional analgesia technique during the entire 72h postoperative period or non receiving the PCA morphine as a rescue analgesia technique will be dropped out from the study for the primary outcome. The primary outcome is the total consumption of morphine during the first three post-operative days. Secondary end points are daily consumption of morphine, pain values at rest and during movement measured with visual analogue scales, QOL 15 analysis at day 3 and at the end of the hospital stay, and specifically the adverse events related to both regional analgesia techniques.

Sample size Considering the study of Kigma and colleagues (ref), the patients receiving a TEA for scopic oesophagectomy reported a MME consumption at 24h 14 mg for the whole 72h postoperative period. We hypothesize no difference (0 mg) between groups (i.e, standard (TEA) group and experimental (ESP) group). The hypothesis is that the amount of morphine needed in the ESP group is not higher but instead similar or less than that in the TEA group. If there is truly no difference between the standard (TEA) and experimental (ESP) treatment, then 25 patients are required with a 80% power (ß risk) for a lower limit of a one-sided 97.5% confidence interval (or equivalently a 95% two-sided confidence interval) to be below the non-inferiority limit of +10 (see table of sample size calculations). Assuming loss of follow-up is approximately 10%, a total of 28 patients are needed for both groups The primary end point will be the total consumption of morphine as rescue analgesia at the end of the first 72 postoperative hours. The T-test will be used to test the non-inferiority comparing the difference (µ2- µ1) to a non-zero quantity M. The assumptions of the t-test are: 1. The data are continuous (not discrete). 2. The differences follow a normal probability distribution. 3. The study sample is a simple random sample from its population. Each individual in the population has an equal probability of being selected in the sample. A Man Whitney test will be used if the data are nonparametric.

For the secondary end points, linear mixed effect models will be used taking into account repeated measures in the same patient (group, time and patient effect), such as for plasma concentration of ropivacaine, the daily amount of Ropivacaine, . Fisher test will be used for the comparison of categorical variables such as adverse events) . Mann Whitney test will be used for the endpoints mentionned above.

Switching to superiority hypothesis If the confidence interval for the difference between both groups (µ2- µ1) lies entirely below 0, then it is acceptable to calculate the P-value associated with a test of superiority and to evaluate whether this is sufficiently small to reject convincingly the hypothesis of no difference. There is no multiplicity argument that affects this interpretation because, in statistical terms, it corresponds to a simple closed test procedure. Usually this demonstration of a benefit is sufficient on its own, provided the safety profiles of the new intervention and the comparator are similar.

All statistical tests are 2 sided with significant level of 0.05. All analysis will be done with latest version of R statistical software. For the first 3 postoperative days, data will be recorded during routine patient rounds done by the anesthesia team in the ICU and surgical ward. Another set of data will be recorded after one month, during routine patient follow-up.

The study will be performed in accordance with the ethical principles that originated from the Declaration of Helsinki, ICH GCP, and all applicable regulations.

Participant Information and Consent A written informed consent shall be obtained from each participant before entering the study or performing any unusual or nonroutine procedure that involves risk to the participant.

Before recruitment and enrollment, each prospective participant or his or her legal guardian will be given a full explanation of the study, allowed to read the approved Information consent form (ICF), and allowed to have any questions answered. Once the investigator is assured that the participant/legal guardian understands the implications of participating in the study, the participant/legal guardian will be asked to give consent to participate in the study by signing the ICF. The authorized person obtaining the informed consent will also sign the ICF.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with esophageal cancer and scheduled to for TLE using Akiyama technique,
* Informed and signed the consent

Exclusion Criteria:

* patient refusal,
* allergy to local anesthetic (LA),
* complex congenital malformation,
* mental deficit,
* substance abuse (alcohol, opioids, etc.)
* renal insufficiency

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Morphine consumption | 72 hours
  mg morphine

SECONDARY OUTCOMES:
Extension of sensory blockade | 72hours
  number of metamere blockade
Side effects | 72hours
  the percentage of patients with at least one of the following adverse events: Hypoblood pressure, Urinary retention, post dural puncture heachache
quality of recovery | 1 week
  QOR 15 from 0 minimal value to 150 maximal value

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Macaire, MD, Principal Investigator — Vinmec Healthcare System

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chan KKW, Saluja R, Delos Santos K, Lien K, Shah K, Cramarossa G, Zhu X, Wong RKS. Neoadjuvant treatments for locally advanced, resectable esophageal cancer: A network meta-analysis. Int J Cancer. 2018 Jul 15;143(2):430-437. doi: 10.1002/ijc.31312. Epub 2018 Mar 8. PMID 29441562
- [Result] Gisbertz SS, Hagens ERC, Ruurda JP, Schneider PM, Tan LJ, Domrachev SA, Hoeppner J, van Berge Henegouwen MI. The evolution of surgical approach for esophageal cancer. Ann N Y Acad Sci. 2018 Dec;1434(1):149-155. doi: 10.1111/nyas.13957. Epub 2018 Sep 7. PMID 30191569
- [Result] Simonnet G, Rivat C. Opioid-induced hyperalgesia: abnormal or normal pain? Neuroreport. 2003 Jan 20;14(1):1-7. doi: 10.1097/00001756-200301200-00001. No abstract available. PMID 12544821
- [Result] Richebe P, Cahana A, Rivat C. Tolerance and opioid-induced hyperalgesia. Is a divorce imminent? Pain. 2012 Aug;153(8):1547-1548. doi: 10.1016/j.pain.2012.05.002. Epub 2012 May 17. No abstract available. PMID 22608577
- [Result] Rivat C, Bollag L, Richebe P. Mechanisms of regional anaesthesia protection against hyperalgesia and pain chronicization. Curr Opin Anaesthesiol. 2013 Oct;26(5):621-5. doi: 10.1097/01.aco.0000432511.08070.de. PMID 23995064
- [Result] Richebe P, Rivat C, Liu SS. Perioperative or postoperative nerve block for preventive analgesia: should we care about the timing of our regional anesthesia? Anesth Analg. 2013 May;116(5):969-970. doi: 10.1213/ANE.0b013e31828843c9. No abstract available. PMID 23606468
- [Result] Richebe P, Capdevila X, Rivat C. Persistent Postsurgical Pain: Pathophysiology and Preventative Pharmacologic Considerations. Anesthesiology. 2018 Sep;129(3):590-607. doi: 10.1097/ALN.0000000000002238. PMID 29738328
- [Result] Richman JM, Liu SS, Courpas G, Wong R, Rowlingson AJ, McGready J, Cohen SR, Wu CL. Does continuous peripheral nerve block provide superior pain control to opioids? A meta-analysis. Anesth Analg. 2006 Jan;102(1):248-57. doi: 10.1213/01.ANE.0000181289.09675.7D. PMID 16368838
- [Result] Ng A, Swanevelder J. Pain relief after thoracotomy: is epidural analgesia the optimal technique? Br J Anaesth. 2007 Feb;98(2):159-62. doi: 10.1093/bja/ael360. No abstract available. PMID 17251209
- [Result] van Boekel RLM, Warle MC, Nielen RGC, Vissers KCP, van der Sande R, Bronkhorst EM, Lerou JGC, Steegers MAH. Relationship Between Postoperative Pain and Overall 30-Day Complications in a Broad Surgical Population: An Observational Study. Ann Surg. 2019 May;269(5):856-865. doi: 10.1097/SLA.0000000000002583. PMID 29135493
- [Result] Humble SR, Dalton AJ, Li L. A systematic review of therapeutic interventions to reduce acute and chronic post-surgical pain after amputation, thoracotomy or mastectomy. Eur J Pain. 2015 Apr;19(4):451-65. doi: 10.1002/ejp.567. Epub 2014 Aug 4. PMID 25088289
- [Result] Rivat C, Ballantyne J. The dark side of opioids in pain management: basic science explains clinical observation. Pain Rep. 2016 Sep 8;1(2):e570. doi: 10.1097/PR9.0000000000000570. eCollection 2016 Aug. PMID 29392193
- [Result] Yibulayin W, Abulizi S, Lv H, Sun W. Minimally invasive oesophagectomy versus open esophagectomy for resectable esophageal cancer: a meta-analysis. World J Surg Oncol. 2016 Dec 8;14(1):304. doi: 10.1186/s12957-016-1062-7. PMID 27927246
- [Result] Biere SS, van Berge Henegouwen MI, Maas KW, Bonavina L, Rosman C, Garcia JR, Gisbertz SS, Klinkenbijl JH, Hollmann MW, de Lange ES, Bonjer HJ, van der Peet DL, Cuesta MA. Minimally invasive versus open oesophagectomy for patients with oesophageal cancer: a multicentre, open-label, randomised controlled trial. Lancet. 2012 May 19;379(9829):1887-92. doi: 10.1016/S0140-6736(12)60516-9. Epub 2012 May 1. PMID 22552194
- [Result] Joshi GP, Bonnet F, Shah R, Wilkinson RC, Camu F, Fischer B, Neugebauer EA, Rawal N, Schug SA, Simanski C, Kehlet H. A systematic review of randomized trials evaluating regional techniques for postthoracotomy analgesia. Anesth Analg. 2008 Sep;107(3):1026-40. doi: 10.1213/01.ane.0000333274.63501.ff. PMID 18713924
- [Result] Visser E, Marsman M, van Rossum PSN, Cheong E, Al-Naimi K, van Klei WA, Ruurda JP, van Hillegersberg R. Postoperative pain management after esophagectomy: a systematic review and meta-analysis. Dis Esophagus. 2017 Oct 1;30(10):1-11. doi: 10.1093/dote/dox052. PMID 28859388
- [Result] Popping DM, Elia N, Van Aken HK, Marret E, Schug SA, Kranke P, Wenk M, Tramer MR. Impact of epidural analgesia on mortality and morbidity after surgery: systematic review and meta-analysis of randomized controlled trials. Ann Surg. 2014 Jun;259(6):1056-67. doi: 10.1097/SLA.0000000000000237. PMID 24096762
- [Result] Cook TM, Counsell D, Wildsmith JA; Royal College of Anaesthetists Third National Audit Project. Major complications of central neuraxial block: report on the Third National Audit Project of the Royal College of Anaesthetists. Br J Anaesth. 2009 Feb;102(2):179-90. doi: 10.1093/bja/aen360. Epub 2009 Jan 12. PMID 19139027
- [Result] Christie IW, McCabe S. Major complications of epidural analgesia after surgery: results of a six-year survey. Anaesthesia. 2007 Apr;62(4):335-41. doi: 10.1111/j.1365-2044.2007.04992.x. PMID 17381568
- [Result] Kooij FO, Schlack WS, Preckel B, Hollmann MW. Does regional analgesia for major surgery improve outcome? Focus on epidural analgesia. Anesth Analg. 2014 Sep;119(3):740-744. doi: 10.1213/ANE.0000000000000245. No abstract available. PMID 25137006
- [Result] Bos EME, Haumann J, de Quelerij M, Vandertop WP, Kalkman CJ, Hollmann MW, Lirk P. Haematoma and abscess after neuraxial anaesthesia: a review of 647 cases. Br J Anaesth. 2018 Apr;120(4):693-704. doi: 10.1016/j.bja.2017.11.105. Epub 2018 Feb 15. PMID 29576110
- [Result] Kingma BF, Visser E, Marsman M, Ruurda JP, van Hillegersberg R. Epidural analgesia after minimally invasive esophagectomy: efficacy and complication profile. Dis Esophagus. 2019 Aug 1;32(8):doy116. doi: 10.1093/dote/doy116. PMID 30561659
- [Result] Hermanides J, Hollmann MW, Stevens MF, Lirk P. Failed epidural: causes and management. Br J Anaesth. 2012 Aug;109(2):144-54. doi: 10.1093/bja/aes214. Epub 2012 Jun 26. PMID 22735301
- [Result] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Result] Macaire P, Ho N, Nguyen T, Nguyen B, Vu V, Quach C, Roques V, Capdevila X. Ultrasound-Guided Continuous Thoracic Erector Spinae Plane Block Within an Enhanced Recovery Program Is Associated with Decreased Opioid Consumption and Improved Patient Postoperative Rehabilitation After Open Cardiac Surgery-A Patient-Matched, Controlled Before-and-After Study. J Cardiothorac Vasc Anesth. 2019 Jun;33(6):1659-1667. doi: 10.1053/j.jvca.2018.11.021. Epub 2018 Nov 19. PMID 30665850
- [Result] Macaire P, Ho N, Nguyen V, Phan Van H, Dinh Nguyen Thien K, Bringuier S, Capdevila X. Bilateral ultrasound-guided thoracic erector spinae plane blocks using a programmed intermittent bolus improve opioid-sparing postoperative analgesia in pediatric patients after open cardiac surgery: a randomized, double-blind, placebo-controlled trial. Reg Anesth Pain Med. 2020 Oct;45(10):805-812. doi: 10.1136/rapm-2020-101496. Epub 2020 Aug 19. PMID 32817407
- [Result] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) Statement: guidelines for reporting observational studies. Int J Surg. 2014 Dec;12(12):1495-9. doi: 10.1016/j.ijsu.2014.07.013. Epub 2014 Jul 18. PMID 25046131
- [Result] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Result] De Cassai A, Tonetti T, Galligioni H, Ori C. [Erector spinae plane block as a multiple catheter technique for open esophagectomy: a case report]. Braz J Anesthesiol. 2019 Jan-Feb;69(1):95-98. doi: 10.1016/j.bjan.2018.06.001. Epub 2018 Nov 17. PMID 30459088
- [Result] Gamble C, Krishan A, Stocken D, Lewis S, Juszczak E, Dore C, Williamson PR, Altman DG, Montgomery A, Lim P, Berlin J, Senn S, Day S, Barbachano Y, Loder E. Guidelines for the Content of Statistical Analysis Plans in Clinical Trials. JAMA. 2017 Dec 19;318(23):2337-2343. doi: 10.1001/jama.2017.18556. PMID 29260229
- See also: PROSPECT Recommendations, Thoracotomy 2015 — https://esraeurope.org/prospect/procedures/thoracotomy